CLINICAL TRIAL: NCT06196749
Title: Clinical Study of the Application of Modified Ultrasound-Guided Dynamic Needle Tip Positioning Technique in Percutaneous Distal Radial Artery Catheterization
Brief Title: Ultrasound-Guided Technique in Distal Radial Artery Catheterization Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Collaborators: Health and Family Planning Commission of Guangdong (Other Government)
Responsible Party: Principal Investigator, Yupeng Liang, Director, Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: B2021044
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Coronary Arteriography; Distal Radial Artery; Percutaneous Coronary Intervention; Ultrasonography, Doppler

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified ultrasound-guided dynamic needle tip positioning technique group (Experimental): Perform distal radial arterial cannulation using modified ultrasound-guided dynamic needle tip positioning technique
  Interventions: Procedure: Perform distal radial arterial cannulation using modified ultrasound-guided dynamic needle tip positioning technique
- Palpation group (Active Comparator): Perform radial arterial cannulation under palpation guidance
  Interventions: Procedure: Palpation guided puncture

INTERVENTIONS:
Procedure: Perform distal radial arterial cannulation using modified ultrasound-guided dynamic needle tip positioning technique — This study employs a modified ultrasound-guided dynamic needle tip positioning technique for distal radial arterial cannulation. The technique uses an ultrasound probe with two wires to create an acoustic shadow, improving needle tip visibility. Real-time dynamic tracking assists in precise needle placement within the distal radial artery through the nose-horn region. This method is used for coronary angiography and potential percutaneous coronary interventions, aiming to increase success rates and reduce complications like hematoma, nerve injury, and arterial spasm, thus enhancing safety and efficiency.
  Arms: Modified ultrasound-guided dynamic needle tip positioning technique group
Procedure: Palpation guided puncture — Perform distal radial arterial cannulation under palpation guidance
  Arms: Palpation group

SUMMARY:
The research project is focused on examining the clinical effectiveness of an enhanced ultrasound dynamic needle tip positioning method for guiding distal radial artery puncture and catheterization. Anticipated results suggest that the improved ultrasound dynamic needle tip positioning method will surpass tactile guidance in terms of the success rate of the first puncture attempt, as well as overall puncture and catheterization success rates.

DETAILED DESCRIPTION:
The distal radial artery access route has several advantages; however, it comes with drawbacks like tortuous anatomy and a smaller lumen diameter. Compared to the wrist radial artery approach, it is more prone to spasm and has a lower success rate for puncture and catheterization. This clinical study aims to explore the effectiveness of an enhanced ultrasound dynamic needle tip positioning method for guiding distal radial artery puncture and catheterization.

In this prospective, randomized, single-center study, we will enroll 112 patients scheduled for percutaneous coronary angiography. They will be randomly assigned to either the control group (56 cases) or the study group (56 cases) using digital odd-even randomization. The control group will undergo conventional tactile guidance, while the study group will be guided by the improved ultrasound dynamic needle tip positioning method.

Parameters to be compared between the two groups include the success rate of the first puncture attempt, overall puncture success rate, number of puncture attempts, success rate of catheterization, time to successful catheterization, proportion of sheath sizes used, incidence of hematoma, and incidence of radial artery occlusion 24 hours post-procedure. The anticipated outcome is that the improved ultrasound dynamic needle tip positioning method will enhance the success rate of the first puncture attempt, overall puncture success rate, and catheterization success rate, while reducing the number of puncture attempts and operation time.

ELIGIBILITY:
Inclusion Criteria:

Patients between the ages of 18 and 85 who agree to undergo coronaroangiography

Exclusion Criteria:

1. Absence of radial artery pulsatility.
2. Abnormal Allen test.
3. Hemodynamic instability.
4. Preoperative ultrasound showing a distal radial artery diameter less than 1.8mm.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
First Needle Puncture Success Rate | Immediately after the puncture procedure
  The proportion of participants who successfully achieve a first puncture into the radial artery on their first attempt.
Puncture success rate | Immediately after the puncture procedure
  The proportion of participants who achieve successful puncture of the radial artery on their attempt
Cannulation Success Rate | Immediately after the cannulation procedure is completed
  The proportion of participants who successfully achieve cannulation of the radial artery after a puncture attempt.

SECONDARY OUTCOMES:
Number of Punctures | Immediately after the puncture procedure
  The total number of puncture attempts required to successfully cannulate the radial artery.
Puncture Success Time | Immediately after the puncture procedure
  The duration of time elapsed from the initiation of the puncture attempt until the successful completion of the puncture.
Distal Radial Hematoma Rate | Immediately after the puncture and again within 24 hours
  The proportion of participants who develop a hematoma at the puncture site on the distal radial artery.
24-Hour Proximal Radial Occlusion Rate | 24 hours after the procedure
  The proportion of participants who experience radial artery occlusion at the proximal site within 24 hours after the procedure.
24-Hour Distal Radial Occlusion Rate | 24 hours after the procedure
  The proportion of participants who experience radial artery occlusion at the distal site within 24 hours after the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Yupeng Liang, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No